CLINICAL TRIAL: NCT01314053
Title: Retrospective Evaluation of Safety and Efficacy of Daptomycin Used in Patients With Serious Gram-positive Infections
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wen-Sen Lee, Department of Infectious Disease, WanFang Hospital
Other Study IDs: 99084
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Serious Gram-positive Infections
Keywords: Daptomycin; Serious Gram-positive Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Daptomycin was approved since 2005 in Taiwan and have been studied and published in west countries. After review the published papers, the few data were described in the Asian countries or Taiwan. The objectives of this study are to evaluate the efficacy and safety of daptomycin for the treatment of Gram-positive infections under actual conditions of use, and to understand other information concerned with daptomycin prescription. This study represents an opportunity for acquiring real world data on daptomycin usage, and may provide physicians in Taiwan with the information of characteristic of the patients receiving daptomycin and to evaluate outcomes. It also provides a means to identify safety signals that emerge with clinical usage.

DETAILED DESCRIPTION:
This is a retrospective, non-comparative study, which will be performed after obtaining permission from the institutional review board. Patients with serious gram-positive infections who had received daptomycin from January 2009 and completed daptomycin therapy by the end of December 2010 will be screened, and patients who received ≥ 3 days of daptomycin will be identified eligible to be included. Eligible patients' medical records will be reviewed.

As this is a retrospective chart review, it is expected that informed consent will not be necessary. For patients' confidentiality concern, patients' name or chart number will not to be record in any part of Data Collection Form (APPENDIX 1). A patient identification number will be assigned to each patient included in this surveillance. A study coordinator at site will be identified, and hospital specific process will be utilized to identify patients. Information to be collected was shown on Data Collection Form (Appendix 1). After completing patient data collection, the efficacy and safety will be evaluated for the included cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients started daptomycin therapy since January 2009.
* Patients completed daptomycin therapy by the end of December 2010.
* Patients had Gram positive infections.
* Patients received daptomycin therapy for at least 3 days.

Exclusion Criteria:

* Daptomycin therapy will be chosen by the treating physician based on clinical indication and it is expected that risks of therapy will have already been considered.
* subjects are only to be excluded if he/she was enrolled in any antibiotics clinical trial during daptomycin treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients who are prescribed daptomycin as part of required medical care for gram positive infections as deemed necessary by his/her treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Study Completion 2011-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Sen Lee, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan